CLINICAL TRIAL: NCT07393022
Title: A Single-Dose, Open-Label, Randomized, Two-Way Crossover, Bioequivalence Study of Levetiracetam 1500 mg Coated Granules in Sachet Formulations (Desitin Arzneimittel GmbH, Germany) and Keppra 2 x 750 mg Film-Coated Tablet Formulations (UCB Pharma, Germany) in Healthy, Male and Non-Pregnant, Non-Lactating Female Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Levetiracetam 1500 mg Coated Granules in Healthy, Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LEV-004/K
Record Dates: First submitted 2025-12-01; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Pharmacokinetic Analysis; Bioequivalence; Health Adult Subjects
Keywords: single dose; randomized; bioequivalence; two-period; crossover; levetiracetam
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Intervention Model Description: randomized, 2-period, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levetiracetam 1500 mg (Experimental): Levetiracetam 1500 mg coated granules, single oral dose
  Interventions: Drug: Levetiracetam 1500 mg
- Keppra 750 mg (Active Comparator): Keppra 750 mg film-coated tablets, single oral dose of two tablets
  Interventions: Drug: Keppra® 750 mg

INTERVENTIONS:
Drug: Levetiracetam 1500 mg — coated granules, single oral dose
  Arms: Levetiracetam 1500 mg
Drug: Keppra® 750 mg — single oral dose of two tablets
  Arms: Keppra 750 mg

SUMMARY:
Pivotal, single-dose, randomized, open-label, two-period, two-sequence, two-treatment, single-centre, crossover, bioequivalence study of Levetiracetam 1500 mg coated granules in sachet formulations and Keppra (Levetiracetam) 2 x 750 mg film-coated tablet formulations in healthy male and female under fasting conditions.

DETAILED DESCRIPTION:
This will be a pivotal, single-dose, randomized, open-label, two-period, two-sequence, two-treatment, single-centre, crossover, bioequivalence study of Levetiracetam 1500 mg coated granules in sachet formulations and Keppra (Levetiracetam) 2 x 750 mg film-coated tablet formulations in healthy, non-smoking, male and non-pregnant, non-lactating female. The products will be studied using a crossover design with 20 healthy, non-smoking, male and non-pregnant, non-lactating female volunteers being administered an oral dose of 1 × 1500 mg coated granules in sachet (Test Drug A) or 2 x 750 mg film-coated tablets (Reference Drug B) under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking (for at least 6 months prior to first drug administration) male and non-pregnant female volunteers, 18 years of age and older, inclusive.
2. BMI that is between 18.5-30.0 kg/m², inclusive.
3. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
4. QTc interval ≤ 450 milliseconds for males and ≤ 470 milliseconds for females, unless deemed otherwise by the PI/Sub-Investigator.
5. Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, and heart rate between 50-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
6. Clinical laboratory values within BPSI's most recent acceptable laboratory test range, and/or values are deemed by the PI/Sub-Investigator as "Not Clinically Significant".
7. Ability to comprehend and be informed of the nature of the study, as assessed by BPSI staff. Capable of giving written informed consent prior to any study- related procedure. Must be able to communicate effectively with clinic staff.
8. Ability to fast for at least 14 hours and consume standard meals.
9. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
10. Agree not to have a tattoo or body piercing until the end of the study.
11. Agree not to drive or operate heavy machinery if feeling dizzy or drowsy following study drug administration until full mental alertness is regained.
12. Female participants must fulfill at least one of the following:

    * Be surgically sterile for a minimum of 6 months (achieved through partial or total hysterectomy, bilateral oophorectomy, bilateral tubal ligation or bilateral salpingectomy); BPSI Protocol Number: 2953 Sponsor Protocol Number: LEV-004/K Protocol Version Number: 1.0, Dated: Oct-14-2025 Levetiracetam 1500 mg coated granules in sachet formulations Fasting Conditions Page 19 of 51
    * Post-menopausal for a minimum of 1 year (postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause), confirmed by FSH test;
    * Agree to avoid pregnancy and use medically acceptable method of contraception from at least 30 days prior to the study until 30 days after the study has ended (last study procedure).

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first study drug administration, as determined by the PI/Sub-Investigator.
3. Estimated creatinine clearance <60 ml/min, unless determined as not clinically significant by the PI/Sub-Investigator.
4. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
5. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
6. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), breath alcohol test and cotinine. Positive pregnancy test for female participants.
7. Known history or presence of:

   * Alcohol abuse or dependence within one year prior to first study drug administration;
   * Drug abuse or dependence;
   * Significant reaction (allergic, anaphylactic, hypersensitivity, angioedema) or severe response to levetiracetam, their excipients and to any other drug or food unless deemed by the PI/Sub-I as "Not Clinically Significant.";
   * Stevens-Johnson syndrome (SJS);
   * Toxic Epidermal Necrolysis (TEN);
   * Drug Reaction with Eosinophilia and Systemic Symptoms (DRESS);
   * Seizure associated with a particular genetic mutation called SCN8A mutation; BPSI Protocol Number: 2953 Sponsor Protocol Number: LEV-004/K Protocol Version Number: 1.0, Dated: Oct-14-2025 Levetiracetam 1500 mg coated granules in sachet formulations Fasting Conditions Page 21 of 51

   Suicidal ideation, attempts and/or behaviour, as assessed by the C-SSRS (baseline version) - Appendix B;

   • Presence of any dietary restrictions unless deemed by the PI/Sub-I as "Not Clinically Significant".
8. Intolerance to and/or difficulty with blood sampling through venipuncture.
9. Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets etc.
10. Individuals who have donated, in the days prior to first study drug administration:

    * 50-499 mL of blood in the previous 30 days;
    * 500 mL of blood or more in the previous 56 days.
11. Donation of plasma by plasmapheresis within 7 days prior to first study drug administration.
12. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first study drug administration.
13. Use of any prescription medication within 14 days prior to first study drug administration (except for medically acceptable contraceptive products).
14. Use of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements) within 14 days prior to first study drug administration (except for medically acceptable contraceptive products).
15. Consumption of food or beverages containing grapefruit and/or pomelo within 10 days prior to first study drug administration.
16. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing in each study period.
17. Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.
18. Difficulty with swallowing whole tablets or granules.
19. Women who are pregnant or lactating.
20. Unable or unwilling to provide informed consent.
21. Have had a tattoo or body piercing within 30 days prior to first study drug administration.

    BPSI Protocol Number: 2953 Sponsor Protocol Number: LEV-004/K Protocol Version Number: 1.0, Dated: Oct-14-2025 Levetiracetam 1500 mg coated granules in sachet formulations Fasting Conditions Page 22 of 51
22. A participant who, in the opinion of the investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence between Levetiracetam Desitin 1500 mg coated granules and Keppra | From enrollment to the end of clinical phase at 2 weeks
  Bioequivalence is concluded under fasting conditions if the 90% confidence interval for the Test/Reference ratios of geometric means for AUCt and Cmax are contained within the ICH-defined acceptance range of 80-125% for levetiracetam
AUC | From enrollment to the end of the study at 1 week
  Area under Curve

CONTACTS AND LOCATIONS:
Locations (1):
- Biopharma Services Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
internal confidential data